CLINICAL TRIAL: NCT02329028
Title: Feasibility of Mini-EEG in the Prehospital Setting
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Johannes Björkman, Resident, Helsinki University Central Hospital
Other Study IDs: 150/13/03/02/2013
Record Dates: First submitted 2014-08-08; First posted 2014-12-31 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Epilepsy; Coma
Keywords: Emergency Care, Prehospital; Electroencephalography; Coma
MeSH Terms: conditions — Epilepsy; Coma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Prehospital mini-EEG: Feasibility of prehospital EEG device in unconscious patients.
  Interventions: Device: Prehospital mini-EEG

INTERVENTIONS:
Device: Prehospital mini-EEG — Observational

SUMMARY:
The EEG is widely used in the diagnosis of central nervous system pathology, including epileptic seizures and epilepsy. Presently, EEG is available only during office hours in most hospitals, pending on the availability of a clinical neurophysiologist and the lack of oncall possibility outside these hours. Standard EEG devices are large and their operation require meticulous application of several leads. The department of clinical neurophysiology at Helsinki University Central Hospital has developed a mini-EEG device for use in the emergency department as well as in the prehospital setting. The aims of this pilot study is to evaluate the feasibility of the mini-EEG in the prehospital setting. Patients with a decreased level of consciousness, as evaluated by the emergency medical provider on the scene, are included. The mini--EEG device is to be used by a specially trained emergency medical supervisor. EEG is otherwise obtained in a normal fashion, but only three electrodes are used. The sample size is 30. Data are collected as a part of the clinical work in daily practice. The aim is to collect observational data on feasibility, no clinical interventions will be performed based on the EEG. No funding is needed as data is collected during daily work.

The mini-EEG is a prototype EEG/EKG-adapter, designed by Helsinki Univeristy Central Hospital, and as such, does not have a trade name. It is to be connected to a monitor/defibrillator used by the EMS personel, currently the LifePak 15, manufactured by Physio-Control, Redmond, WA 98052. (www.physio-control.com)

ELIGIBILITY:
Inclusion Criteria:

* Unconsciousness resulting in activation of the local EMS units

Exclusion Criteria:

* Cardiac arrest
* Traumatic unconsciousness
* Transient unconsciousness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unconscious patients in the prehospital field
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2015-01; Primary Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Signal interpretability | 60 min
  evaluated by a physician (ex 0=unworthy, 1=interfered, 2=good quality)
Device ease-of-use | 60 min
  evaluated by ems field staff (0=not fit for field use ....... 5=optimal for field use)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Silfvast, MD, Ph.D, Study Director — Helsinki University Central Hospital; Tapani Salmi, MD, Ph.D., Study Director — Helsinki University Central Hospital; Johannes Björkman, MD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland